CLINICAL TRIAL: NCT07259551
Title: Effect of the Palming Technique on Preoperative Anxiety and Hemodynamic Responses in Thyroid Surgery
Status: Completed | Type: Observational
Sponsor: Yuzuncu Yil University (Other)
Responsible Party: Principal Investigator, Nureddin YUZKAT, Associate professor, Yuzuncu Yil University
Other Study IDs: The Palming Technique
Record Dates: First submitted 2025-11-15; First posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2022-02

CONDITIONS: Preoperative Anxiety and Associated Hemodynamic Changes
Keywords: Hemodynamics; intubation; preoperative anxiety; relaxation techniques; thyroidectomy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group P: Patients who received the palm-based technique
  Interventions: Behavioral: Group P
- Group N: Control group without intervention

INTERVENTIONS:
Behavioral: Group P — When admitted to the preoperative waiting room (T1), all patients:
  Baseline vital signs (SpO₂, heart rate, blood pressure) State-Trait Anxiety Inventory (STAI) scores were recorded. Patients in Group P received the palm-based technique; Group N received no intervention.
  The same parameters were measured again 15 minutes later (T2).
  After transfer to the operating room, standard monitoring was performed, and hemodynamic data were recorded at the following times:
  Pre-intubation (T3)
  1 min (T4), 3 min (T5), 5 min (T6), and 10 min (T7) after intubation Main Outcome Measures: Changes in preoperative anxiety level Changes in hemodynamic parameters after the palmar technique
  Groups: Group P

SUMMARY:
Purpose of the Observational Study: The purpose of this observational study was to evaluate the effects of the palmar technique on preoperative anxiety, hemodynamic parameters, and intubation-related hemodynamic responses in patients undergoing thyroidectomy.

Primary Research Question: Does the palmar technique applied preoperatively reduce preoperative anxiety and associated hemodynamic changes in thyroidectomy patients? Study Design: Type: Prospective, single-blind, observational study Location: A single-center tertiary care hospital in Turkey Sample: 80 patients aged 18-65, ASA I-II

Methods:

Patients were divided into two groups using a sealed envelope method:

Group P: Patients who received the palm-based technique Group N: Control group without intervention

When admitted to the preoperative waiting room (T1), all patients:

Baseline vital signs (SpO₂, heart rate, blood pressure) State-Trait Anxiety Inventory (STAI) scores were recorded. Patients in Group P received the palm-based technique; Group N received no intervention.

The same parameters were measured again 15 minutes later (T2).

After transfer to the operating room, standard monitoring was performed, and hemodynamic data were recorded at the following times:

Pre-intubation (T3)

1 min (T4), 3 min (T5), 5 min (T6), and 10 min (T7) after intubation Main Outcome Measures: Changes in preoperative anxiety level Changes in hemodynamic parameters after the palmar technique Sample Size:Total: 80 patients

DETAILED DESCRIPTION:
Purpose of the Observational Study: The purpose of this observational study was to evaluate the effects of the palmar technique on preoperative anxiety, hemodynamic parameters, and intubation-related hemodynamic responses in patients undergoing thyroidectomy.

Primary Research Question: Does the palmar technique applied preoperatively reduce preoperative anxiety and associated hemodynamic changes in thyroidectomy patients? Study Design: Type: Prospective, single-blind, observational study Location: A single-center tertiary care hospital in Turkey Sample: 80 patients aged 18-65, ASA I-II

Methods:

Patients were divided into two groups using a sealed envelope method:

Group P: Patients who received the palm-based technique Group N: Control group without intervention

When admitted to the preoperative waiting room (T1), all patients:

Baseline vital signs (SpO₂, heart rate, blood pressure) State-Trait Anxiety Inventory (STAI) scores were recorded. Patients in Group P received the palm-based technique; Group N received no intervention.

The same parameters were measured again 15 minutes later (T2).

After transfer to the operating room, standard monitoring was performed, and hemodynamic data were recorded at the following times:

Pre-intubation (T3)

1 min (T4), 3 min (T5), 5 min (T6), and 10 min (T7) after intubation Main Outcome Measures: Changes in preoperative anxiety level Changes in hemodynamic parameters after the palmar technique Sample Size:Total: 80 patients

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-65 years
* Patients classified as ASA I-II
* Patients scheduled for thyroid surgery
* Patients without a history of glaucoma
* Patients without active psychiatric or neurological disease
* Patients who were informed about the study and provided written informed consent

Exclusion Criteria:

* Patients with a diagnosed psychiatric disorder
* Patients using sedatives, antidepressants, or antiepileptic medications
* Patients with impaired cooperation, comprehension, vision, or hearing
* Patients with a history of ophthalmic surgery
* Patients classified as ASA III or higher

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consisted of adult patients scheduled to undergo thyroidectomy at a tertiary care hospital in Türkiye. A total of 80 patients aged 18-65 years and classified as ASA I-II according to the American Society of Anesthesiologists physical status classification were included. All participants were thoroughly informed about the study procedures and provided written informed consent. Eligible patients had no active psychiatric or neurological disorders, no history of glaucoma, and no prior ophthalmic surgery. Following randomization, patients were assigned to either the palming group (n = 40) or the control group (n = 40).
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-04-15 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
Change in Preoperative Anxiety Score (State-Trait Anxiety Inventory - STAI-State) | Baseline (T1) and 15 minutes after intervention (T2)
  Baseline (TPreoperative anxiety will be assessed using the State-Trait Anxiety Inventory - State (STAI-State) scale (range: 20-80; higher scores indicate higher anxiety). The primary outcome is the change in STAI-State score from baseline (T1) to 15 minutes after the palming technique (T2).1) and 15 minutes after intervention (T2)
Change in Heart Rate | Baseline (T1) and 15 minutes after intervention (T2)
  Change in heart rate (beats per minute) between baseline (T1) and 15 minutes after the palming technique (T2).

CONTACTS AND LOCATIONS:
Overall Officials: Nureddin Yuzkat, Principal Investigator — Yuzuncu Yil University
Locations (1):
- Van Yüzüncü Yıl Universitesi, Van, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be made available to other researchers due to confidentiality considerations and because data sharing was not included in the informed consent obtained from participants.

REFERENCES:
- [Background] Wang R, Huang X, Wang Y, Akbari M. Non-pharmacologic Approaches in Preoperative Anxiety, a Comprehensive Review. Front Public Health. 2022 Apr 11;10:854673. doi: 10.3389/fpubh.2022.854673. eCollection 2022. PMID 35480569
- See also: Bates method. In: Wikipedia [Internet]. 2025 [cited 2025 May 11]. — https://en.wikipedia.org/w/index.php?title=Bates_method&oldid=1289654741